CLINICAL TRIAL: NCT04295031
Title: AMEMET Study - Observational Multicentric Clinical Study: Metformin in Patients Over 65 Years With Type 2 Diabetes (DM2)
Brief Title: Metformin in Older Adults With Type 2 Diabetes (AMEMET)
Acronym: AMEMET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Associazione Medici Endocrinologi (Other)
Responsible Party: Sponsor
Other Study IDs: AMEMET Study
Record Dates: First submitted 2020-02-21; First posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DM2 without renal disease: patients with type 2 diabetes with normal renal function
- DM2 with renal impairment: patients with type 2 diabetes with impaired renal function

SUMMARY:
Multicentric, observational, cross-sectional study in Italy. The aims are to evaluate the daily metformin prescribed dose and the impact of renal function and concomitant medication in diabetic patients over 65 years.

DETAILED DESCRIPTION:
The study was commissioned by the Italian Association of Clinical Endocrinologists (Association of Medical Endocrinologists - AME) and approved by the Ethical Committee of Cuneo Hospital. The research was open to all specialists taking care of patients with diabetes in Italy.

The primary endpoint was the evaluation of metformin dosage. Secondary endpoints were the relationship between the metformin dosage and the renal filtration rate and the relationship between the metformin dosage and the concomitant medication.

An ad hoc form was developed and used to record all medical findings. The form was emailed to all participating centers who then emailed or faxed it back to the investigator's data manager. Data were checked for accuracy.

The following data were required: age, gender, body weight and height, diabetes duration, type of metformin (classical/slow), daily dosage of metformin, reported side effects,concomitant medications.

Serum creatinine and HbA1c levels obtained within the previous two months were also required.

Each participating center recruited about 50 diabetic outpatients. Inclusion criteria were as follows: adult outpatients ≥ 65 years with T2 diabetes mellitus, using metformin for at least six months, usually assuming three daily meals, and capable of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* adult outpatients (≥65 years);
* T2 diabetes mellitus;
* Taking metformin for at least six months;
* assuming three daily meals;
* capable of informed consent.

Exclusion Criteria:

* severe liver or renal failure (eGFR <30 mL/min/1.73 m2);
* hospitalization for any cause in the last six month;
* glucocorticoid treatment in the last six month;
* oncologic treatment in the last six month;
* Ramadan in the last six months.

Ages: 65 Years to 90 Years | Sex: All
Age Groups: Older Adult
Study Population: All diabetic patients respecting eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
metformin daily dose in diabetic outpatients type 2 | six months
  relationship between metformin dose and filtration rate

SECONDARY OUTCOMES:
renal filtration rate | six months
  relationship between metformin rate and concomitant medication

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Borretta, MD, Principal Investigator — Associazione Medici Endocrinologi
Locations (1):
- AME - Associazione Medici Endocrinologi, Udine, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] LeRoith D, Biessels GJ, Braithwaite SS, Casanueva FF, Draznin B, Halter JB, Hirsch IB, McDonnell ME, Molitch ME, Murad MH, Sinclair AJ. Treatment of Diabetes in Older Adults: An Endocrine Society* Clinical Practice Guideline. J Clin Endocrinol Metab. 2019 May 1;104(5):1520-1574. doi: 10.1210/jc.2019-00198. PMID 30903688
- [Result] Davies MJ, D'Alessio DA, Fradkin J, Kernan WN, Mathieu C, Mingrone G, Rossing P, Tsapas A, Wexler DJ, Buse JB. Management of hyperglycaemia in type 2 diabetes, 2018. A consensus report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2018 Dec;61(12):2461-2498. doi: 10.1007/s00125-018-4729-5. PMID 30288571
- [Result] Garber AJ, Abrahamson MJ, Barzilay JI, Blonde L, Bloomgarden ZT, Bush MA, Dagogo-Jack S, DeFronzo RA, Einhorn D, Fonseca VA, Garber JR, Garvey WT, Grunberger G, Handelsman Y, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Rosenblit PD, Umpierrez GE. CONSENSUS STATEMENT BY THE AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY ON THE COMPREHENSIVE TYPE 2 DIABETES MANAGEMENT ALGORITHM - 2019 EXECUTIVE SUMMARY. Endocr Pract. 2019 Jan;25(1):69-100. doi: 10.4158/CS-2018-0535. No abstract available. PMID 30742570
- [Result] Schlender L, Martinez YV, Adeniji C, Reeves D, Faller B, Sommerauer C, Al Qur'an T, Woodham A, Kunnamo I, Sonnichsen A, Renom-Guiteras A. Efficacy and safety of metformin in the management of type 2 diabetes mellitus in older adults: a systematic review for the development of recommendations to reduce potentially inappropriate prescribing. BMC Geriatr. 2017 Oct 16;17(Suppl 1):227. doi: 10.1186/s12877-017-0574-5. PMID 29047344